CLINICAL TRIAL: NCT02264665
Title: AN OBSERVATIONAL REAL-WORLD STUDY OF THE SYSTEMIC TREATMENT OF WELL-DIFFERENTIATED, UNRESECTABLE OR METASTATIC, PROGRESSIVE PANCREATIC NEUROENDOCRINE TUMOURS (PNET): A STUDY OF MORBIDITY AND MORTALITY AT 2 YEARS
Brief Title: OPALINE : A Study Of Morbidity And Mortality At 2 Years
Acronym: OPALINE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Novartis (Industry); Keyrus Biopharma (Other)
Responsible Party: Sponsor
Other Study IDs: A6181214; OPALINE (Other: Alias Study Number)
Record Dates: First submitted 2014-09-02; First posted 2014-10-15 (Estimated); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Neuroendocrine Tumor, Well Differentiated and Progressive
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Sunitinib; Everolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sunitinib
  Interventions: Drug: sunitinib
- Afinitor
  Interventions: Drug: everolimus
- other treatment (chémotherapy, SSA..)
  Interventions: Drug: chemotherapies recommended in france

INTERVENTIONS:
Drug: sunitinib — sunitinib 37.5mg/d orally
  Groups: Sunitinib
Drug: everolimus — everolimus 10mg/d orally
  Groups: Afinitor
Drug: chemotherapies recommended in france — depends on the chemotherapy prescribed (IV)
  Groups: other treatment (chémotherapy, SSA..)

SUMMARY:
A descriptive, prospective (partly retrospective), multisite, observational study conducted in France in adult patients treated for a well differentiated, unresectable or metastatic, pancreatic neuroendocrine tumor with disease progression.

DETAILED DESCRIPTION:
prospective and retrospective Analyses will be performed using SAS® software

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age;
* Patients treated with a targeted therapy (sunitinib, everolimus) or with other treatments (interferon, or metabolic radiotherapy, or chemotherapy or somatostatin analog)* for:

  *Patients whose treatment line (targeted therapy or other treatment) is initiated as a 1st, 2nd, 3rd or 4th line of therapy at the time of inclusion (incident patients) or patients receiving their 1st, 2nd, 3rd or 4th line of therapy provided that treatment was initiated in the site in which the patient is enrolled in the study (prevalent patients); a change of line is defined as a change in molecule or combination.
* A histologically confirmed unresectable or metastatic pancreatic neuroendocrine tumor;
* Well-differentiated;
* Progressive prior to initiation of treatment in the investigator's judgment (clinical or radiological progression);
* Patients who have been informed of the conditions of the study and who have signed the informed consent.

Exclusion Criteria:

* Patients with a diagnosis of poorly differentiated neuroendocrine carcinoma or an adenoneuroendocrine carcinoma.
* Patients receiving targeted therapy (everolimus or sunitinib) already received in a previous line of treatment (rechallenged patient).
* Patients refusing to give consent.
* Patients receiving a fifth line or subsequent line of systemic treatment.
* Patients participating in a clinical trial in a treatment arm not validated by the MA and the TNCD according to the version dated December 2013.
* Patients randomized to the placebo arm of a placebo-controlled trial or to a double-blind trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with progressive, metastatic or unresectable, and well differentiated pancreatic neuroendocrine tumors
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- France (35):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - Hopital Saint-Andre, Bordeaux
  - CHU de Caen, Caen
  - Cabinet Medical, Challes-les-Eaux
  - CHRU de Tours - Hôpital TROUSSEAU, Chambray-lès-Tours
  - Hopital d'Estaing, Clermont-Ferrand
  - Hopital du Bocage, Dijon
  - Unite d'Oncologie Digestive, Departement d'HGE, Grenoble
  - Centre Oscar Lambret, Lille
  - Chu Dupuytren Service Oncologie, Limoges
  - CH Bretagne Sud, Lorient
  - Hopital Edouard Herriot - Pavillon H - Service d'oncologie digestive, Lyon
  - Hopital Edouard Herriot - Service d'Oncologie Digestive, Pavillon H, Lyon
  - Hopital Edouard Herriot, Pavillion O, Oncologie Medicale, Lyon
  - Hopital La Timone Service de Gastroenterologie et Oncologie Digestive, Marseille
  - CHR d'Annecy, Metz-Tessy
  - Centre Val D'Aurelle-Paul Lamarque, Montpellier
  - CRLC Val d'Aurelle, Montpellier
  - Hopital de LA Source, Centre Hospitalier Regional, Orléans
  - CH Pitie Salpetriere, Paris
  - Hopital Cochin, Paris
  - Groupe Hospitalier Cochin, Paris
  - Hopital Saint Jean, Perpignan
  - Hôpital Haut Lévèque, Pessac
  - Hopital de Cornouaille, Quimper
  - C.H.U. de Reims - Hôpital Robert Debré, Reims
  - Hopital Robert Debre, Service D'Hepato-gastro-enterolo, Reims
  - Clinique Armoricaine, Saint-Brieuc
  - Pôle Hospitalier Mutualiste, Saint-Nazaire
  - Clinique Mutualiste de l'estuaire, Saint-Nazaire
  - CHU de Strasbourg - Hopital de Hautepierre / Service de Medecine Interne et Nutrition, Strasbourg
  - Hopital Foch, Onco Hermatologie, Suresnes
  - Cabinet Medical, Vannes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Smith D, Lepage C, Vicaut E, Dominguez S, Coriat R, Dubreuil O, Lecomte T, Baudin E, Venat Bouvet L, Samalin E, Santos A, Borie O, Bisot-Locard S, Goichot B, Lombard-Bohas C. Observational Study in a Real-World Setting of Targeted Therapy in the Systemic Treatment of Progressive Unresectable or Metastatic Well-Differentiated Pancreatic Neuroendocrine Tumors (pNETs) in France: OPALINE Study. Adv Ther. 2022 Jun;39(6):2731-2748. doi: 10.1007/s12325-022-02103-7. Epub 2022 Apr 13. PMID 35419649
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181214&StudyName=Observational%20Study%20In%20Real%20Life%20Settings%20Of%20The%20Systemic%20Treatment%20Of%20Well%20Differentiated%2C%20Unresectable%20Or%20Metastatic%2C%20Progressive%20Panc

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational study carried out in France in adult participants treated for a well-differentiated, unresectable or metastatic, progressive pancreatic neuroendocrine tumor (pNET).
Groups:
- Everolimus (Targeted Therapy) at Inclusion: Participants included in this reporting group were those who at the time of inclusion in the study either initiated treatment with everolimus or were being treated with everolimus. Participants were prospectively followed-up for 2 years in this study.
- Sunitinib (Targeted Therapy) at Inclusion: Participants included in this reporting group were those who at the time of inclusion in the study either initiated treatment with sunitinib or were being treated with sunitinib. Participants were prospectively followed-up for 2 years in this study.
- Chemotherapy (Other Treatment) at Inclusion: Participants included in this reporting group were those who at the time of inclusion in the study either initiated treatment with chemotherapy or were being treated with chemotherapy. Participants were prospectively followed-up for 2 years in this study.
- Somatostatin Analogues (Other Treatment) at Inclusion: Participants included in this reporting group were those who at the time of inclusion in the study either initiated treatment with somatostatin analogues or were being treated with somatostatin analogues. Participants were prospectively followed-up for 2 years in this study.
- Metabolic Radiotherapy (Other Treatment) at Inclusion: Participants included in this reporting group were those who at the time of inclusion in the study either initiated treatment with metabolic radiotherapy or were being treated with metabolic radiotherapy. Participants were prospectively followed-up for 2 years in this study.
- Interferon-alpha (Other Treatment) at Inclusion: Participants included in this reporting group were those who at the time of inclusion in the study either initiated treatment with interferon-alpha or were being treated with interferon-alpha. Participants were prospectively followed-up for 2 years in this study.
- Treatment Not Documented: This reporting group consisted of those participants whose treatment was not documented at time of inclusion.
Period: Overall Study
Arm/Group | Everolimus (Targeted Therapy) at Inclusion | Sunitinib (Targeted Therapy) at Inclusion | Chemotherapy (Other Treatment) at Inclusion | Somatostatin Analogues (Other Treatment) at Inclusion | Metabolic Radiotherapy (Other Treatment) at Inclusion | Interferon-alpha (Other Treatment) at Inclusion | Treatment Not Documented
Started | 35 | 23 | 52 | 30 | 1 | 0 | 3
Reference Set (Full Analysis Set) | 32 | 23 | 50 | 28 | 1 | 0 | 0
Safety Set | 35 | 23 | 52 | 30 | 1 | 0 | 0
Completed | 22 | 15 | 31 | 21 | 1 | 0 | 0
Not Completed | 13 | 8 | 21 | 9 | 0 | 0 | 3
Not completed — Other | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Death | 9 | 8 | 13 | 5 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Participant decision | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Inclusion/non-inclusion criteria not respected | 3 | 0 | 2 | 2 | 0 | 0 | 2
Not completed — Data Missing | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis (FAS) (reference) set included participants who met the eligibility criteria and had received at least 1 dose of the treatment documented during the prospective follow-up period (the treatment start date must be completed and the treatment stop date must be after the date of inclusion if the start date is prior to the date of inclusion) in the study (targeted therapy or other treatment) and excluded the participants with no follow-up data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus (Targeted Therapy) at Inclusion | Sunitinib (Targeted Therapy) at Inclusion | Chemotherapy (Other Treatment) at Inclusion | Somatostatin Analogues (Other Treatment) at Inclusion | Metabolic Radiotherapy (Other Treatment) at Inclusion | Total
Number analyzed (Participants) | 32 | 23 | 50 | 28 | 1 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.16 (12.56) | 64.19 (12.27) | 62.06 (12.39) | 66.77 (12.76) | 82.38 | 63.35 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 5 | 18 | 11 | 1 | 53
  Male | 14 | 18 | 32 | 17 | 0 | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) at 2 Years Assessed by Investigator Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 - Based on Type of Treatment at Inclusion
Description: PFS was defined as time (in months) from date of start of treatment (the treatment line ongoing at the time of inclusion in the study) to first documentation of disease progression (PD) or date of death due to any cause, when receiving the main treatment at the time of inclusion. RECIST v1.1, PD: at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study treatment (this included baseline sum if that is smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). Unequivocal progression of existing non-target lesions. Appearance of 1 or more new target or non-target lesions. If a participant did not have an event, data censoring was done at the last recorded time to PD or the last tumor assessment, last disease assessment. Analysis was performed using Kaplan-Meier method.
Time Frame: At 2 years of prospective follow-up
Population: FAS included participants who met eligibility criteria, received at least 1 dose of treatment during prospective follow-up period (treatment start date must be completed, treatment stop date must be after date of inclusion if start date is prior to date of inclusion) in the study (targeted therapy or other treatment) and excluded participants with no follow-up data. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus (Targeted Therapy) at Inclusion | Sunitinib (Targeted Therapy) at Inclusion | Chemotherapy (Other Treatment) at Inclusion | Somatostatin Analogues (Other Treatment) at Inclusion | Metabolic Radiotherapy (Other Treatment) at Inclusion
Number analyzed (Participants) | 32 | 23 | 50 | 27 | 1
Percentage of participants | 26.5 [10.3 to 46.0] | 19.3 [4.6 to 41.4] | 36.5 [13.8 to 60.0] | 38.6 [16.0 to 61.0] | NA [NA to NA] — Survival analysis not performed with only one participant at risk.

2. Primary Outcome: PFS at 2 Years Assessed by Investigator Per RECIST v1.1 - Based on Targeted Therapy Group and Other Treatments Group at Inclusion
Description: PFS was defined as time (in months) from date of start of treatment (the treatment line ongoing at the time of inclusion in the study) to first documentation of PD or date of death due to any cause, when receiving the main treatment at the time of inclusion. RECIST v1.1, PD: at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study treatment (this included baseline sum if that is smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. Appearance of 1 or more new target or non-target lesions. If a participant did not have an event, data censoring was done at the last recorded time to PD or the last tumor assessment, last disease assessment. Analysis was performed using Kaplan-Meier method.
Time Frame: At 2 years of prospective follow-up
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Targeted Therapy at Inclusion: Participants included in this reporting group were those who at the time of inclusion in the study either initiated treatment with targeted therapies or were being treated with targeted therapies. Participants were prospectively followed-up for 2 years in this study.
- Other Treatments at Inclusion: Participants included in this reporting group were those who at the time of inclusion in the study either initiated treatment with other treatments or were being treated with other treatments. Participants were prospectively followed-up for 2 years in this study.
Arm/Group | Targeted Therapy at Inclusion | Other Treatments at Inclusion
Number analyzed (Participants) | 55 | 78
Percentage of participants | 19.9 [9.2 to 33.4] | 29.0 [14.7 to 45.0]

3. Primary Outcome: Overall Survival (OS) Rate at 2 Years - Based on Type of Treatment at Inclusion
Description: OS was the percentage of participants who were alive at 2 years of prospective follow-up. OS was defined as the time (in months) from the date of start of treatment (of the treatment line ongoing at the time of inclusion in the study) to the date of death due to any cause. Participants with no event or lost to follow-up or alive at the end of the study were censored at their last follow-up date (last follow-up date or last news). Analysis was performed using Kaplan-Meier method.
Time Frame: At 2 years of prospective follow-up
Population: FAS included participants who met eligibility criteria, received at least 1 dose of treatment during prospective follow-up period (treatment start date must be completed, treatment stop date must be after date of inclusion if start date is prior to date of inclusion) in the study (targeted therapy or other treatment) and excluded participants with no follow-up data. Here, "Overall Number of Participants" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus (Targeted Therapy) at Inclusion | Sunitinib (Targeted Therapy) at Inclusion | Chemotherapy (Other Treatment) at Inclusion | Somatostatin Analogues (Other Treatment) at Inclusion | Metabolic Radiotherapy (Other Treatment) at Inclusion
Number analyzed (Participants) | 32 | 23 | 50 | 28 | 1
Percentage of participants | 60.2 [37.6 to 76.8] | 68.4 [37.8 to 86.2] | 69.6 [52.6 to 81.6] | 79.7 [48.0 to 93.2] | NA [NA to NA] — Survival analysis not performed with only one participant at risk.

4. Primary Outcome: OS Rate at 2 Years- Based on Targeted Therapy Group and Other Treatments Group at Inclusion
Description: as for outcome 3
Time Frame: At 2 years of prospective follow-up
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Targeted Therapy at Inclusion | Other Treatments at Inclusion
Number analyzed (Participants) | 55 | 79
Percentage of participants | 63.9 [46.8 to 76.8] | 71.7 [57.2 to 82.1]

5. Primary Outcome: Number of Participants With Reasons for Temporary and Permanent Treatment Discontinuation - Based on Targeted Therapy Group and Other Treatment Group at Inclusion
Time Frame: During 2 years of prospective follow-up
Population: Safety analysis set included participants who received at least one dose of the documented treatment in the study (targeted therapy or other treatment). If the participant was prevalent, the treatment must still be ongoing at the time of inclusion in the study and if the participant was incident, the treatment must be started at or after inclusion in the study. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Therapy at Inclusion | Other Treatments at Inclusion
Number analyzed (Participants) | 20 | 22
Participants
  Adverse event | 12 | 6
  Doctor's choice | 1 | 11
  Participant's choice | 3 | 3
  Other | 4 | 2

6. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment Related AEs, SAEs and SAEs With Common Terminology Criteria For Adverse Events (CTCAE) 3, 4 and 5, v4.0-Based on Treatment Received At-least Once During Study
Description: AE: any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. SAE: any AE, regardless of dose, that: led to death; was life-threatening; required hospitalization or prolonged hospitalization; led to persistent or significant incapacity or led to congenital anomaly or birth defect. Treatment-related AE was any untoward medical occurrence attributed to study drug in participant who received study drug. Relatedness to treatment was assessed by investigator. Per CTCAE 4.0, Grade 3 (Severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4=Life-threatening events Grade 5 (Death) events=death related to an AE. Participants in this outcome measure were grouped according to type of treatment received at least once during study irrespective of treatment they initiated or were receiving at time of inclusion.
Time Frame: During 2 years of prospective follow-up
Population: Safety analysis set. Since participants were grouped on the basis of type of treatment they received at least once during 2 years of follow-up, participants are not exclusive per treatment arm. One participant could have received more than 1 type of treatment during these 2 years.
Measure: Count of Participants; unit: Participants
Groups:
- Everolimus During Study: Participants who received everolimus at least once in the study.
- Sunitinib During Study: Participants who received sunitinib at least once in the study.
- Chemotherapy During Study: Participants who received chemotherapy at least once in the study.
- Somatostatin Analogues During Study: Participants who received somatostatin analogues at least once in the study.
- Metabolic Radiotherapy During Study: Participants who received metabolic radiotherapy at least once in the study.
- Other Than Study Treatments During Study: Participants who received treatment other than the study treatments at least once in the study.
Arm/Group | Everolimus During Study | Sunitinib During Study | Chemotherapy During Study | Somatostatin Analogues During Study | Metabolic Radiotherapy During Study | Other Than Study Treatments During Study
Number analyzed (Participants) | 52 | 36 | 82 | 65 | 11 | 16
Participants
  AE | 43 | 32 | 63 | 48 | 6 | 8
  Treatment Related AE | 31 | 24 | 48 | 13 | 2 | 0
  SAE | 21 | 9 | 26 | 24 | 3 | 3
  Treatment Related SAE | 6 | 2 | 5 | 1 | 1 | 0
  At least one grade 3 AE | 21 | 11 | 18 | 14 | 1 | 3
  At least one grade 3 SAE | 14 | 6 | 12 | 12 | 0 | 0
  At least one AE of grade 4 or higher | 6 | 2 | 18 | 16 | 2 | 1

7. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation of Treatment - Based on Treatment Received At-least Once During the Study
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Participants in this outcome measure were grouped according to type of treatment received at least once during study irrespective of treatment they initiated or were receiving at time of inclusion.
Time Frame: During 2 years of prospective follow-up
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Somatostatin Analogues During Study at Inclusion: Participants who received somatostatin analogues at least once in the study.
- Other Than Study Treatment During Study: Participants who received treatment other than the study treatments at least once in the study.
Arm/Group | Everolimus During Study | Sunitinib During Study | Chemotherapy During Study | Somatostatin Analogues During Study at Inclusion | Metabolic Radiotherapy During Study | Other Than Study Treatment During Study
Number analyzed (Participants) | 52 | 36 | 82 | 65 | 11 | 16
Participants
  Temporary discontinuation of treatment | 15 | 9 | 11 | 8 | 0 | 1
  Permanent discontinuation of treatment | 14 | 10 | 12 | 12 | 0 | 1

8. Primary Outcome: Number of Participants With Adverse Events Leading to Death - Based on Treatment Received At-least Once During the Study
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Adverse events leading to death are reported in this outcome measure. Participants in this outcome measure were grouped according to type of treatment received at least once during study irrespective of treatment they initiated or were receiving at time of inclusion.
Time Frame: During 2 years of prospective follow-up
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus During Study | Sunitinib During Study | Chemotherapy During Study | Somatostatin Analogues During Study at Inclusion | Metabolic Radiotherapy During Study | Other Than Study Treatments During Study
Number analyzed (Participants) | 52 | 36 | 82 | 65 | 11 | 16
Participants | 3 | 2 | 11 | 12 | 2 | 1

9. Secondary Outcome: Mean of Number of Tumor Assessment Visits - Based on Targeted Therapy Group and Other Treatments Group at Inclusion
Time Frame: During 2 years of prospective follow-up
Population: FAS included participants who met eligibility criteria, received at least 1 dose of treatment during prospective follow-up period (treatment start date must be completed, treatment stop date must be after date of inclusion if start date is prior to date of inclusion) in the study (targeted therapy or other treatment) and excluded participants with no follow-up data.
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Targeted Therapy at Inclusion | Other Treatments at Inclusion
Number analyzed (Participants) | 55 | 79
Visits | 5.8 (2.7) | 5.5 (2.7)

10. Secondary Outcome: Number of Participants According to Frequency of Tumor Assessment Visits - Based on Targeted Therapy Group and Other Treatments Group at Inclusion
Description: Frequency = number of tumor assessment visits /([last visit date - baseline date]/365.25).
Time Frame: During 2 years of prospective follow-up
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Therapy at Inclusion | Other Treatments at Inclusion
Number analyzed (Participants) | 55 | 79
Participants
  0 tests per annum | 2 | 3
  2 tests per annum | 3 | 4
  3 tests per annum | 19 | 26
  4 tests per annum | 18 | 30
  5 tests per annum | 10 | 10
  6 tests per annum | 2 | 4
  7 tests per annum | 1 | 0
  9 tests per annum | 0 | 2

11. Secondary Outcome: Number of Participants With Different Types of Investigation Used for Tumor Assessment - Based on Targeted Therapy Group and Other Treatments Group at Inclusion
Description: The different types of investigations were performed for assessment of tumor regardless of treatment received. Investigations performed were Computed Tomography (CT) scan, Magnetic Resonance Imaging (MRI), Positron Emission Tomography (PET) scan, Octreoscan, Ultrasound. All the investigations were used at least once during the study for all treatments.
Time Frame: During 2 years of prospective follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Therapy at Inclusion | Other Treatments at Inclusion
Number analyzed (Participants) | 53 | 76
Participants
  CT Scan | 48 | 65
  MRI | 28 | 45
  PET Scan | 11 | 15
  Octreoscan | 13 | 15
  Ultrasound | 6 | 4
  Imaging (CT scan and/or MRI) | 52 | 74

12. Secondary Outcome: Number of Participants Who Had a Change in Their Treatment - Based on Targeted Therapy Group and Other Treatments Group at Inclusion
Description: In this outcome measure, number of participants with a change in treatment compared to treatment at inclusion is reported.
Time Frame: During 2 years of prospective follow-up
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Therapy at Inclusion | Other Treatments at Inclusion
Number analyzed (Participants) | 55 | 79
Participants | 44 | 68

13. Secondary Outcome: Number of Participants According to Number of Changes in Doses of Treatment - Based on Type of Treatment (Everolimus, Sunitinib, Chemotherapy and Somatostatin Analogues) at Inclusion
Description: Number of participants according to number of changes in doses of treatment is reported for this outcome measure.
Time Frame: During 2 years of prospective follow-up
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus (Targeted Therapy) at Inclusion | Sunitinib (Targeted Therapy) at Inclusion | Chemotherapy (Other Treatment) at Inclusion | Somatostatin Analogues (Other Treatment) at Inclusion
Number analyzed (Participants) | 32 | 23 | 50 | 28
Participants
  0 | 25 | 18 | 40 | 21
  1 | 4 | 3 | 7 | 7
  2 | 1 | 2 | 3 | 0
  4 | 2 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants According to Course of Changes in Doses of Treatment - Based on Type of Treatment (Metabolic Radiotherapy) at Inclusion
Description: Number of participants according to course of changes in doses of treatment is reported for this outcome measure.
Time Frame: During 2 years of prospective follow-up
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Metabolic Radiotherapy (Other Treatment) at Inclusion
Number analyzed (Participants) | 1
Participants
  0 | 0
  1 | 0
  2 | 0
  4 | 1

15. Secondary Outcome: Number of Combined Main Lines of Treatments Received - Based on Targeted Therapy Group and Other Treatments Group at Inclusion
Description: The number of lines of combined main treatment administered during the study were assessed.
Time Frame: During 2 years of prospective follow-up
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Treatment lines
Arm/Group | Targeted Therapy at Inclusion | Other Treatments at Inclusion
Number analyzed (Participants) | 55 | 79
Treatment lines | 3.9 (1.7) | 2.9 (1.6)

16. Secondary Outcome: Number of Main Lines of Treatment Received During the Study - Based on Targeted Therapy Group and Other Treatments Group at Inclusion
Description: The number of main lines of treatment received during the study treatment are reported in this outcome measure.
Time Frame: During 2 years of prospective follow-up
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Treatment lines
Arm/Group | Targeted Therapy at Inclusion | Other Treatments at Inclusion
Number analyzed (Participants) | 55 | 79
Treatment lines | 3.7 (1.7) | 2.8 (1.5)

17. Secondary Outcome: Number of Participants With Types of Main Lines of Treatment Received During the Follow-up - Based on Targeted Therapy Group and Other Treatments Group at Inclusion
Description: The types of main lines of treatment included 1st line, 2nd line, 3rd line, 4th line, 5th line, 6th line, 7th line and 8th line.
Time Frame: During 2 years of prospective follow-up
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Therapy at Inclusion | Other Treatments at Inclusion
Number analyzed (Participants) | 55 | 79
Participants
  1st line | 8 | 38
  2nd line | 27 | 43
  3rd line | 25 | 30
  4th line | 28 | 26
  5th line | 15 | 15
  6th line | 7 | 2
  7th line | 4 | 1
  8th line | 2 | 0

ADVERSE EVENTS:
Time Frame: During 2 years of prospective follow-up
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Participants during course of study changed their treatment, irrespective of treatment at the time of inclusion. Safety data reported is according to treatment taken at least once during the study.
Arm/Group | Everolimus During Study | Sunitinib During Study | Chemotherapy During Study | Somatostatin Analogues During Study | Metabolic Radiotherapy During Study | Other Than Study Treatment During Study
All-Cause Mortality (participants affected / at risk) | 4/52 | 3/36 | 15/82 | 14/65 | 2/11 | 1/16
Serious Adverse Events (participants affected / at risk) | 21/52 | 9/36 | 26/82 | 24/65 | 3/11 | 3/16
Other Adverse Events (participants affected / at risk) | 39/52 | 29/36 | 56/82 | 41/65 | 4/11 | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus During Study (N=52) | Sunitinib During Study (N=36) | Chemotherapy During Study (N=82) | Somatostatin Analogues During Study (N=65) | Metabolic Radiotherapy During Study (N=11) | Other Than Study Treatment During Study (N=16)
Disease progression (General disorders) | 3 | 2 | 5 | 8 | 0 | 1
General physical health deterioration (General disorders) | 4 | 0 | 4 | 4 | 0 | 0
Condition aggravated (General disorders) | 0 | 0 | 2 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 — Reasons for death were unknown for both the participants.
Pyrexia (General disorders) | 2 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 0 | 1 | 0 | 0
Oedema (General disorders) | 1 | 1 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Gastric varices (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Prostatitis Escherichia coli (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 2 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 2 | 0 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus During Study (N=52) | Sunitinib During Study (N=36) | Chemotherapy During Study (N=82) | Somatostatin Analogues During Study (N=65) | Metabolic Radiotherapy During Study (N=11) | Other Than Study Treatment During Study (N=16)
Asthenia (General disorders) | 5 | 6 | 24 | 8 | 1 | 2
Mucosal inflammation (General disorders) | 8 | 3 | 2 | 3 | 0 | 0
Oedema peripheral (General disorders) | 5 | 1 | 3 | 3 | 0 | 2
Pyrexia (General disorders) | 4 | 2 | 4 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 1 | 1 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 4 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 1 | 1
Oedema (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 0
Device related thrombosis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Drug intolerance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 9 | 12 | 11 | 2 | 3
Nausea (Gastrointestinal disorders) | 4 | 0 | 14 | 4 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4 | 7 | 3 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 5 | 2 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 6 | 2 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4 | 3 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 3 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 5 | 3 | 5 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 9 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 6 | 2 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 1 | 1 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Psychomotor skills impaired (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 8 | 7 | 3 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 10 | 3 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 3 | 4 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Macrocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0
Folliculitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Dermatophytosis of nail (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 3 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 3 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2 | 0 | 0
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 6 | 4 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0 | 0
Cell death (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 3 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hair disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 4 | 2 | 2 | 3 | 0 | 3
Blood phosphorus decreased (Investigations) | 0 | 3 | 2 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 1 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood calcium abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood sodium abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Gammaglutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Prothrombin time ratio decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pericardial disease (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Nail injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Persistent corneal epithelial defect (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 2 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 1 | 1 | 0 | 1
Cholangitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depressive symptom (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Liver transplant (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT02264665/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT02264665/SAP_001.pdf